CLINICAL TRIAL: NCT02413073
Title: Effectiveness of Whole Body Vibration for Patients With Chronic Kidney Disease in the Interdialytic Period on Muscle Strength, Balance, Quality of Life and Functional Capacity: Randomized Clinical Trial
Brief Title: Whole Body Vibration in Kidney Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Helen Fisio, Principal Investigator, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 35872014.8.00005208
Record Dates: First submitted 2014-11-29; First posted 2015-04-09 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Kidney Disease
Keywords: whole body vibration; kidney disease
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham of Whole Body Vibration (Sham Comparator): This group will receive placebo treatment on the platform we'll use a little engine that will produce a very small vibration stimulus in the platform.
  Interventions: Procedure: Whole Body Vibration
- Whole body vibration Group (Experimental): This group will be a training na vibratory platform with 12 weeks (3 months), held twice a week on alternate days
  Interventions: Procedure: Whole Body Vibration

INTERVENTIONS:
Procedure: Whole Body Vibration — We wil use vibration in patients with kidney disease

SUMMARY:
There are no studies in the literature evaluating the vibration of the whole body in patients with chronic renal failure. The study aims to assess the effectiveness of whole body vibration in patients with renal disease in the final phase in the interdialytic period. It will be a randomized, triple-blind, controlled and randomized. The pilot study will be 20 individuals initially. In intervention patients will be randomly divided into two groups: sham platform and platform. As a result it is expected that the training of whole body vibration may promote patient compliance, since it requires less physical effort for implementation and greater comfort in the application, thus allowing the sedentary and / or less active patients can benefit by to minimize the harmful effects of physical inactivity associated with pre-existing kidney problems.

DETAILED DESCRIPTION:
Studies of chronic kidney disease has conventional hemodialysis and physical therapy exercises as the most relevant interventions in the treatment and maintenance of the quality of life of these patients, but recent studies have shown significant results also in training with whole body vibration, especially for muscle strengthening, balance and quality of life of patients with different diseases. However, there are no studies in the literature analyzing whole-body vibration in patients with chronic renal failure.

Objective: To evaluate the effectiveness of wholy body vibration in patients with renal disease in the final stage in the interdialytic period.

Materials and Methods: A clinical trial randomized, triple-blind (patient, appraiser and statistics) controlled and supplied with random distribution. The study will be conducted in Cardiopulmonary Therapy Physical Therapy Laboratory of the Federal University of Pernambuco (UFPE). The sample is calculated from a pilot study to be carried out previously. The pilot study will be 20 subjects, 10 patients in each of the two groups.

In intervention patients will be randomly assigned to one of two groups: platform and platform sham. Training twice a week for 3 consecutive months. The evaluations will be conducted in two periods: before and after the intervention. The assessment tools are included: the isokinetic dynamometer to evaluate the maximal voluntary isometric contraction of the knee extensors, the Biodex Balance System to evaluate the static and dynamic body balance, the quality of life questionnaire specific for Chronic Renal patient - Kidney Disease Quality of Life - short Form (KDQOL-SFTM), and the 6-minute walk test to assess the functional capacity of the patient.

Expected results: It is expected that training in vibrating platform can promote patient compliance, since it requires less physical effort for implementation and greater comfort in the application, thus allowing the sedentary patients and / or less active can benefit , thus minimizing the harmful effects of physical inactivity associated with pre-existing kidney problems.

ELIGIBILITY:
Inclusion criteria:

* Patients diagnosed with kidney disease, of both sexes, aged between 18 and 65 and on hemodialysis program for at least 3 months without the osteomusculoesquelético system changes that hamper the tests.

Exclusion criteria:

* Patients who heart failure, hypertension and uncontrolled arrhythmias, metal implants, pregnancy, thrombosis history, stroke sequelae.

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-04; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
muscle strength, as measured by isokinetic dynamometer (Kgf) | 3 months

SECONDARY OUTCOMES:
postural equilibrium, as measured by biodex balance (score) | 3 months
functional capacity, as measured by 6MWT | 3 months
quality of life, as measured by questionnaire | 3 months
Thickness of Quadriceps Muscle, as measured by ultrasound | 3 mounths

CONTACTS AND LOCATIONS:
Overall Officials: Helen KB Fuzari, MD, Principal Investigator — Universidade Federal de Pernambuco